CLINICAL TRIAL: NCT01813513
Title: A Phase I, Randomized, Multiple-Dose Study to Evaluate the Pharmacokinetic Drug-Drug Interaction Between IDX719 and Simeprevir in Healthy Subjects
Brief Title: Study to Evaluate Drug-Drug Interaction Between IDX719 and Simeprevir in Healthy Participants (MK-1894-004)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1894-004; IDX-06A-004 (Other: Idenix Protocol Number)
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Hepatitis C Infection
Keywords: HCV; Hepatitis C Virus; Hepatitis C; antiviral drugs; liver
MeSH Terms: conditions — Hepatitis C | interventions — samatasvir; Simeprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A: IDX719 then IDX719/Simeprevir (Experimental): Healthy participants take IDX719 150 mg once daily (QD) on Days 1-7 and IDX719 150 mg QD + simeprevir 150 mg QD on Days 8-14.
  Interventions: Drug: IDX719; Drug: Simeprevir
- Group B: Simeprevir then IDX719/Simeprevir (Experimental): Healthy participants take simeprevir 150 mg QD on Days 1-7 and IDX719 150 mg QD + simeprevir 150 mg QD on Days 8-14.
  Interventions: Drug: IDX719; Drug: Simeprevir
- Group C: IDX719 (Experimental): Healthy participants take IDX719 150 mg QD on Days 1-14.
  Interventions: Drug: IDX719
- Group D: IDX719/Simeprevir (Experimental): Participants from Groups A and B will be asked to return for Group D. Participants take IDX719 and simeprevir QD on Days 1-7 to determine the impact of food on single-dose (on Day 1) and steady state (Day 7) PK.
  Interventions: Drug: IDX719; Drug: Simeprevir
- Group E: High-Fat then Low-Fat PK (Experimental): Participants from Group C will return to determine the PK of IDX719 after high-fat (Day 1) and low-fat (Day 7) meals (Days 2-6 are drug-free washout).
  Interventions: Drug: IDX719
- Group F: Low-Fat then High-Fat PK (Experimental): Participants from Group C will return to determine the PK of IDX719 after low-fat (Day 1) and high-fat (Day 7) meals (Days 2-6 are drug-free washout).
  Interventions: Drug: IDX719

INTERVENTIONS:
Drug: IDX719 — 50 mg tablet for oral administration
  Other Names: Samatasvir
Drug: Simeprevir — 150 mg capsule for oral administration
  Other Names: Olysio™
  Arms: Group A: IDX719 then IDX719/Simeprevir; Group B: Simeprevir then IDX719/Simeprevir; Group D: IDX719/Simeprevir

SUMMARY:
The purpose of this 3-part study is to evaluate the potential impact of simeprevir and food on pharmacokinetics (PK) of IDX719 in healthy participants. Part 1 will evaluate potential PK interactions between IDX719 and simeprevir. Part 2 will evaluate the effect of food on the PK of IDX719 in combination with simeprevir. Part 3 will evaluate the impact of high- versus low-fat meals on the PK of IDX719.

ELIGIBILITY:
Inclusion Criteria:

* Has no clinically significant abnormalities on medical history, physical examination, or 12-lead electrocardiogram (ECG)
* Agrees to use a double method of birth control (one of which must be a barrier) from Screening through at least 90 days after the last dose of study drug
* Agrees to avoid nicotine-containing products from 3 months prior to Screening and for the duration of the study

Exclusion Criteria:

* Is positive for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, or anti-human immunodeficiency virus (HIV) antibodies
* Is pregnant or breastfeeding
* Has previously received either IDX719 or simeprevir
* Has participated in another clinical drug study within 30 days of Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) at steady-state over dosing interval (AUCss) | Up to 30 days
Maximum observed plasma concentration (Cmax) | Up to 30 days
AUC from time zero to infinity | Up to 30 days
Trough plasma concentration (Ctrough) | Up to 30 days

SECONDARY OUTCOMES:
Percentage of participants experiencing serious adverse events (SAEs) | Up to 30 days
Percentage of participants experiencing adverse events (AEs) | Up to 30 days
Percentage of participants experiencing Grade 1-4 laboratory abnormalities | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC